CLINICAL TRIAL: NCT04843748
Title: Clinical Study for Assessing the Visual Performance of Hanita Lenses New Trifocal Intraocular Lens
Brief Title: Clinical Evaluation Study for Assessing the Visual Performance of Hanita Lenses Trifocal IOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hanita Lenses (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HTF-01
Record Dates: First submitted 2021-03-09; First posted 2021-04-14 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-03

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Experimental): single arm open label study
  Interventions: Device: cataract surgery and intraocular lens implantation - both eyes

INTERVENTIONS:
Device: cataract surgery and intraocular lens implantation - both eyes — cataract surgery and intraocular lens implantation for both eyes

SUMMARY:
Hanita Lenses Trifocal IOL, SeeLens AFR (Intensity IOL).Prospective, single-arm single-center, open-label study.

DETAILED DESCRIPTION:
Device: Hanita Lenses Trifocal IOL, SeeLens AFR (Intensity IOL). Indication studied: The Hanita Lenses Trifocal IOL is intended for implantation in the capsular bag in the posterior chamber in order to replace the crystalline lens of the eye to attain visual correction of aphakia in adult patients in whom a cataractous lens has been removed, who desire improved uncorrected vision, useful near and intermediate visual functions, and reduced spectacle dependence.

Study description: This study is a prospective, single-arm single-center, open-label study.

ELIGIBILITY:
Inclusion Criteria:

* Age over 45 years and under 75 years.
* Patients with bilateral age-related cataracts, require bilateral cataract phacoemulsification combined Intraocular Lens implantation;
* Patients with an axial length of 22-24.5mm.
* Normal corneas with less than 0.75D of regular corneal astigmatism.
* Post-operative best-corrected visual acuity projected to be 0.3 logMAR or lower.
* Patient motivated for trifocal IOL after screening by the surgeon.
* Fundus visualization is possible.
* Absence of retinal or optic nerve diseases
* Signed informed consent

Exclusion Criteria:

* Previous ocular/corneal surgery that may affect refraction accuracy or visual acuity.
* Capsule or zonular abnormalities that may affect postoperative centration or tilt of the lens (e.g. pseudoexfoliation syndrome, chronic Uveitis, Marfan's syndrome)
* History or evidence of any ocular disease that may affect visual acuity (i.e. uncontrolled glaucoma, ocular injury, corneal pathologies, retinal pathologies in general and macular pathologies in particular, diabetic retinopathy, uveitis, aniridia or iris atrophy, vitreous pathologies (patients with vitreous separation or floaters can be included).
* Rubella cataract.
* Amblyopia
* Any other ocular condition that may predispose a subject to future complications or contraindicate implantation of the trifocal lens.
* Pupil abnormalities (non-reactive, tonic pupils, abnormally shaped pupils, or pupils that do not dilate at least 3.5 mm under mesopic/scotopic conditions)
* Patients with pupil diameter greater than 4mm in photopic conditions.
* Pregnant, lactating or planning to become pregnant during the course of the trial.
* Allergy or intolerance to required study medications (including antibiotic).
* Subjects participating in a concurrent clinical trial or if they have participated in an ophthalmology clinical trial within the last 30 days.
* Traumatic cataract.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-08-18 (Actual); Primary Completion 2021-01-06 (Actual); Study Completion 2021-01-06 (Actual)

PRIMARY OUTCOMES:
Binocular visual acuity for far, intermediate and near distance after Trifocal IOL implantation | 90-110 days post op
  Binocular visual acuity for far, intermediate and near distance after Trifocal IOL implantation

SECONDARY OUTCOMES:
Defocus Curve | 90-110 days post op
  Will be obtained using an ETDRS chart or PV numbers. Patient's pupil diameter will be evaluated.
  In the statistical stage patients will be categorized according to smaller than 2.5mm, between 2.5 and 4.5mm and above 4.5mm for mesopic and photopic conditions.
  The test will be performed using a phoropter to create defocus in 0.5D increments, starting from 1D to -4D relative to emmetropia so that the patient will be corrected for far vision.
Contrast Sensitivity | 90-110 days post op
  Will be evaluated using a sine wave gratings chart (FACT) at mesopic and photopic conditions. Measurements will be performed with optimal refractive correction.
  Luminance for photopic conditions will be 85cd/m² and 5cd/m² for mesopic conditions. Small deviations are allowed. The working interval for photopic conditions is 75-95cd/m² and for mesopic conditions is 5-15cd/m².
  Luminance for photopic and mesopic conditions will be monitored using Illuminance meter and documented. Results will be expressed as values.
patient satisfaction | 90-110 days post op
  Subjective evaluation will be performed using the modified VF-14 questionnaire for quality of life, in addition to satisfaction questionnaire.

OTHER OUTCOMES:
OCULAR AND INTRAOCULAR BIOMETRICAL MEASUREMENTS | pre- op
  Patients will be examined pre operatively for inclusion and exclusion criteria as well as at the post-operative follow ups for the measurements specified in the flow chart (Section 8.12). These include a validated biometry (Tomey AO-2000, IOL-Master, Lenstar), corneal topography, tomography (optional, performed in accordance with investigator's discretion, retinal OCT, tonometry, slit lamp examination and fundoscopy.
Slit Lamp Exam | 90-110 days post op
  The slit lamp exam will include the measurement of aqueous cell and flare, and the measurement of corneal edema by a standard grading system. It will also include an evaluation for the presence of pupillary irregularities, iris atrophy and pigment dispersion.
  For the evaluation of aqueous cells and flare, use a slit lamp beam 0.3 mm wide and 1 mm high, and use the following grading:
  Cells none (0) = no cells seen trace (+1) = 1-5 cells seen mild (+2) = 6-15 cells seen moderate (+3) = 16-30 cells seen severe (+4) = > 30 cells seen
  Flare none (0) = No Tyndall effect trace (+1) = Tyndall effect barely discernible mild (+2) = Tyndall beam in anterior chamber is mildly intense moderate (+3) = Tyndall beam in anterior chamber is moderately intense severe (+4) = Tyndall beam is severely intense. The aqueous has a white and milky appearance.
VISUAL ACUITY | 90-110 days post op
  Will be measured using an ETDRS chart or PV numbers for distance and PV Numbers Near Vision Card (Precision Vision) for near (40cm) and intermediate distances (80cm). All results will be expressed in logMAR. Visual acuity will be measured in photopic conditions. Monocular BCVA will be measured under mesopic conditions in the follow up of one and three months. NOTE: All charts used should be calibrated to the specific distance to be used during the testing. For example, if the testing distance is 4m, the chart should be calibrated to that distance.

CONTACTS AND LOCATIONS:
Locations (1):
- MeirMC, Kfar Saba, Israel